CLINICAL TRIAL: NCT00063856
Title: A Comparison of Dressing Preparations for Smallpox Vaccination Sites With a Focus Upon the Risk of Secondary Transmission of Vaccinia Virus
Brief Title: Dressing Preparations for Smallpox
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-044
Record Dates: First submitted 2003-07-07; First posted 2003-07-08 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2007-05

CONDITIONS: Smallpox
Keywords: Smallpox, wetvax
MeSH Terms: conditions — Smallpox

INTERVENTIONS:
Biological: Wetvax (APSV)

SUMMARY:
The primary purpose of this study is to find out the risk of spreading the vaccine virus, vaccinia, from the smallpox vaccination site when different types of bandages are used to cover the site. The study will also look at how each bandage type affects the healing of the sore. Study participants will include healthy individuals, 18-50 years old, who have not previously received a smallpox vaccine and healthy individuals, 18-50 years old, who have received a previous smallpox vaccine. All participants will receive the smallpox vaccine and be randomly assigned to 1 of 3 different bandage groups to cover the vaccine site: standard gauze dressing attached with paper tape, Opsite gauze-impregnanted occlusive dressing (attached by paper tape and waterproof), and Allevyn hydropolymer dressing (which is self-adhesive and highly absorbent). Volunteers will be involved in study related procedures for up to 252 days.

DETAILED DESCRIPTION:
This study will investigate the potential for secondary transmission of vaccinia from smallpox vaccination sites covered by various types of dressings, as well as the effects of each dressing type on the healing of the vaccination lesion. The results could have great implications for infection control and public health in the wake of potential mass smallpox vaccination. The study population will consist of two cohorts: healthy individuals who are naive to the smallpox vaccine ("naive group") and healthy individuals who have had previous vaccination with the smallpox vaccine ("experienced group"). Individuals in each group will be vaccinated with a dose of smallpox vaccine diluted to 1:5 and will be randomized to receive one of three dressing preparations to cover the vaccination site: standard 2 inch x 2 inch gauze attached to the skin via paper tape ("Gauze dressing"); Opsite gauze-impregnated occlusive dressing ("occlusive dressing"); and Allevyn hydropolymer dressing (Smith and Nephew, "hydropolymer dressing"). In addition, 30 of the 108 subjects (15 naïve and 15 experienced) will be enrolled as a "cardiac subgroup" and will have additional blood drawn for the assessment of specific biochemical markers related to thrombosis and platelet activation (specifically, plasminogen-activator inhibitor type 1 (PAI-1) and soluble CD40 ligand (sCD40L). The primary study objective will be the assessment of infectivity of vaccination sites via evaluation of vaccinia growth from specimens of the outer dressing for each bandage type. Positive culture reflects failure of the bandage to prevent possible spread of vaccinia. Secondary study objectives include the following: assessment of infectivity of vaccination sites via evaluation of vaccinia growth from specimens from the hand contralateral to the vaccine site for each dressing type; comparison of the rate of lesion healing (time from vaccination until lesion is deemed "well-healed") for each dressing cohort; association of adverse events (AEs) involved with transmission of vaccinia, such as autoinoculation and secondary dissemination, with the type of dressing covering the vaccination site; and determination of the alterations after smallpox vaccination in the body's endogenous fibrinolytic system to investigate the potential pathophysiology of adverse ischemic cardiac events seen in vaccinated subjects in the recent civilian and military campaigns. The tertiary objectives of the study include: assessment of the overall safety profile in each cohort, as determined by reactogenicity of the vaccine and the development of expected and unexpected AEs unrelated to dressing type; assessment of the efficacy of a 1:5 dilution of APSV in vaccinia-experienced adults as measured by the proportion of individuals who respond to vaccination with a "take: 6-11 days after vaccination; characterization of the humoral immune response generated following vaccination in each cohort; assessment of pharyngeal carriage and shedding of vaccinia virus in each cohort of vaccinated volunteers; and assessment of the tolerability of the dressing and total number of bandage changes determined from a volunteer questionnaire and summarized by bandage type. Volunteers will be followed for 56 days following their primary vaccination. Volunteers who do not have a "take" will be offered revaccination under a separate protocol after their 56-day blood sample is drawn. All volunteers will be contacted by telephone for information about serious adverse events at or about 180 days after their primary vaccination.

ELIGIBILITY:
Inclusion Criteria:

A. Vaccinia-naÏve Cohort:

1. Age: 18-32 (children are excluded due to concerns of safety, including autoinoculation).
2. Willing to sign informed consent.
3. Availability for follow-up for planned duration of the study (at least 8 weeks after vaccination).
4. Acceptable medical history by screening evaluation and brief clinical assessment.
5. Absence of a typical vaccinia scar and negative history of smallpox vaccination.
6. Negative serum pregnancy test at screening and negative urine or serum pregnancy test within 24 hours prior to vaccination for woman of childbearing potential. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized.
7. If the volunteer is female and of childbearing potential, she agrees to use acceptable contraception, and not become pregnant for 56 days post vaccination. (Acceptable contraception methods are restricted to effective intrauterine devices (IUDs) or licensed hormonal methods (pills, patch, infection, ring or implant) with use of method for a minimum of 30 days prior to vaccination.)
8. Negative ELISA for HIV or indeterminate Western blot or other assay confirming that the serostatus does not reflect HIV infection.
9. Negative hepatitis B surface antigen and negative antibody to hepatitis C virus.
10. Negative urine glucose by dipstick.
11. ALT <1.5 times institutional upper limit of normal.
12. Adequate renal function defined as a serum creatinine < = 1.5 mg/dl; urine protein < 100 mg/dl or trace or negative proteinuria (by dipstick), and a calculated creatinine clearance >55 mL/min. Formula for calculation is contained within the Manual of Procedures. (Note: Renal function is measured to ensure that subjects could meet criteria for use of cidofovir if needed.)
13. Hematocrit > 34% for females, > 38% for males, platelets > 150,000, WBC > 2,500 and < 11, 000/dL.

B. Vaccinia-experienced Cohort:

1. Evidence of previous receipt of smallpox vaccine before 1989 (via immunization records documenting vaccination or the presence of a typical vaccinia scar).
2. Age 33 to < 50 years.
3. All inclusion criteria used for the vaccinia-naïve cohort, except age and absence of scar or negative history of vaccination.

Exclusion Criteria:

A. Vaccinia-naïve Cohort:

1. History of immunodeficiency.
2. History of myocardial infarction or other ischemic heart disease, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor.
3. The presence on screening ECG of signs suggestive of prior ischemia disease (e.g. Q-waves).
4. The presence of diabetes mellitus.
5. History of an immediate family member (father, mother, brother or sister) who has had onset of ischemic heart disease before age 50 years.
6. Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool. (a) Volunteers ages 18 to < 20 will not need to have this risk assessed, as the tool is predictive only for those age 20 or older.
7. Known or suspectecd impairment of immunologic function including, but not limited to, clinically significant liver disease, moderate to severe kidney impairment.
8. History of or current malignancy except squamous cell or basal cell skin cancer.
9. Active autoimmune disease.
10. Use of immunosuppressive medication (Corticosteroid nasal sprays and inhalers are permissible).
11. History of solid organ or bone marrow transplantation.
12. Medical or psychiatric condition or occupational responsibilities that might preclude subject compliance with the protocol.
13. History of illegal injection drug use.
14. Inactivated vaccine 14 days prior to vaccination.
15. Live attenuated vaccines within 60 days of study.
16. Use of investigational agents under IND within 30 days prior to study.
17. Any history of vaccination with any vaccinia vectored or other pox vectored experimental vaccine.
18. Typical vaccinia scar or history of vaccination.
19. Receipt of blood products or immunoglobulin in the past 6 months.
20. Recent donation of the equivalent of a pint of blood within the 30 days prior to enrollment.
21. Acute febrile illness ( > = 100.5°F) on the day of vaccination.
22. Pregnant or lactating woman.
23. Known IgA deficiency (by history)
24. Eczema of any degree or history of eczema.
25. History of exfoliative skin disorders/conditions. Any acute skin disorders of large magnitude (e.g., laceration requiring sutures, burn greater that 2 x 2 cm).
26. Household contacts/sexual contacts with, or frequent and/or prolonged exposure to, any of the following: (a) pregnant women (b)children < 12 months of age (c) people with eczema or history of eczema (d) people with any of the above skin disorders/conditions (e) people with immunodeficiency disease or use of immunosuppressive medications
27. Health care workers with close contact to individuals with any of the noted excluding underlying illnesses noted above (e.g., HIV+ patients, transplant recipients, patients with eczema).
28. Any condition that, in the opinion of the investigator, might interfere with study objectives.
29. Allergies to any component of the vaccine (e.g., phenol, glycerin, or brilliant green)
30. Allergies to any known component of the diluent.
31. Allergies to any known component of VIG (e.g., thimerosal) or previous allergic reaction to immunoglobulins.
32. Allergies to cidofovir or probenecid.

B. Vaccinia-experienced Cohort:

1. Lack of confirmaton of prior smallpox vaccination.
2. Participation in recent trials (within the last 5 years) of smallpox vaccine.
3. All exclusion criteria used for the vaccinia-naïve cohort except "any history of vaccination with any vaccinia vectored or other pox-vectored experimental vaccine and typical scar or history of vaccination."

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2003-07; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States